CLINICAL TRIAL: NCT02280616
Title: Double-blind, Double-dummy, Randomized, Placebo-controlled, Phase IIa Study on the Efficacy and Tolerability of a 14-day Treatment With Budesonide Effervescent Tablets vs. Viscous Budesonide Suspension vs. Placebo in Patients With Eosinophilic Esophagitis
Brief Title: Budesonide Effervescent Tablets vs. Viscous Budesonide Suspension vs. Placebo in Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUU-2/EEA; 2009-016692-29 (EudraCT Number)
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Budesonide; DNER protein, human; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose budesonide tablet (Experimental)
  Interventions: Drug: low dose budesonide tablet
- High dose budesonide tablet (Experimental)
  Interventions: Drug: high dose budesonide tablet
- High dose budesonide suspension (Experimental)
  Interventions: Drug: high dose budesonide suspension
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: low dose budesonide tablet — 1mg budesonide tablet twice daily AND 5ml placebo suspension twice daily
  Other Names: BET 1mg BID
  Arms: Low dose budesonide tablet
Drug: high dose budesonide tablet — 2mg budesonide tablet twice daily AND 5ml placebo suspension twice daily
  Other Names: BET 2mg BID
  Arms: High dose budesonide tablet
Drug: high dose budesonide suspension — placebo tablet twice daily AND 5ml [0.4mg budesonide/ml] suspension twice daily
  Other Names: BVS 2mg BID
  Arms: High dose budesonide suspension
Drug: Placebo — placebo tablet twice daily AND 5ml placebo suspension twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of a low and high dose of a budesonide effervescent tablet and oral viscous budesonide suspension vs. placebo for the induction treatment of active eosinophilic esophagitis.

ELIGIBILITY:
Major Inclusion Criteria:

* Signed informed consent
* Male or female patients, 18 to 75 years of age
* Confirmed clinicopathological diagnosis of EoE according to established diagnostic criteria:

(A) Clinical symptoms of esophageal dysfunction (B) Peak eosinophils ≥ 15 in at least 1 high-power field (hpf)

- Active symptomatic and histological EoE at baseline

Major Exclusion Criteria:

* Clinically and endoscopically suspicion for gastroesophageal reflux disease, achalasia, or sklerodermia
* Gastroesophageal reflux disease and PPI-responsive esophageal eosinophilia
* Other clinical evident causes than EoE for esophageal eosinophilia
* Any concomitant esophageal disease and relevant gastro-intestinal disease (celiac disease, inflammatory bowel disease, oropharyngeal or esophageal bacterial, viral, or fungal infection)
* Any relevant systemic disease (e.g., AIDS, active tuberculosis)
* Abnormal hepatic function at screening visit, liver cirrhosis, or portal hypertension
* Abnormal renal function at screening
* History of cancer in the last five years (except for non-metastatic cancers, e.g., basalioma)
* History of esophageal surgery at any time or of esophageal dilation procedures within the last 8 weeks prior to screening visit
* Upper gastrointestinal bleeding within 8 weeks prior to screening visit
* Concomitant, or within the 4 weeks prior to screening visit, treatment with systemic therapies for any reason that may affect assessment of primary and secondary endpoints, i.e., systemic glucocorticoids, histamine antagonists, mast cell stabilizers, leukotriene receptor antagonists, biologics, or immunosuppressants
* Concomitant, or within the 2 weeks prior to screening visit, treatment with topical therapies for any reason that may affect assessment of primary and secondary endpoints, i.e., topical glucocorticoids or inhaled sodium cromoglycate
* Installation of dietary restrictions within 4 weeks prior to screening visit or during treatment
* Intake of grapefruit containing food or beverages during the treatment with study medication
* Known intolerance/hypersensitivity to study drug
* Existing or intended pregnancy or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Rate of histological remission | 2 weeks (LOCF)
Change in the mean numbers of eos | 2 weeks (LOCF)

SECONDARY OUTCOMES:
Change in the mean numbers of eos | 2 weeks (LOCF)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mueller, PhD, Study Director — Dr. Falk Pharma GmbH
Locations (1):
- Center for Digestive Diseases Eppendorf, Hamburg, Germany

REFERENCES:
- [Result] Miehlke S, Hruz P, Vieth M, Bussmann C, von Arnim U, Bajbouj M, Schlag C, Madisch A, Fibbe C, Wittenburg H, Allescher HD, Reinshagen M, Schubert S, Tack J, Muller M, Krummenerl P, Arts J, Mueller R, Dilger K, Greinwald R, Straumann A. A randomised, double-blind trial comparing budesonide formulations and dosages for short-term treatment of eosinophilic oesophagitis. Gut. 2016 Mar;65(3):390-9. doi: 10.1136/gutjnl-2014-308815. Epub 2015 Mar 19. PMID 25792708